CLINICAL TRIAL: NCT04829136
Title: Feasibility of Implementing Sustained Oral Fiber Supplementation for Patients Undergoing Allogeneic Hematopoietic Cell Transplantation for Hematological Malignancies
Brief Title: Sustained Oral Fiber Supplementation for Patients Undergoing Donor Stem Cell Transplantation for Hematological Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1121363; NCI-2021-00842 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10599 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-02-26; First posted 2021-04-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm
MeSH Terms: interventions — Parenteral Nutrition; Parenteral Nutrition, Total; Dietary Supplements; Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (enteral nutrition) [Discontinued in January 2024] (Experimental): Patients receive enteral nutrition via nasoenteric feeding tube starting on day 1 until hospital discharge.
  Interventions: Dietary Supplement: Kate Farms 1.0; Other: Survey Administration
- Arm II (standard of care) [Discontinued in January 2024] (Active Comparator): Patients receive standard of care nutritional support.
  Interventions: Dietary Supplement: Standard of Care Nutritional Support; Other: Survey Administration
- Supportive care (Fiber) [Current study activity] (Experimental): Patients receive fiber supplementation PO or enterally starting 14 to 5 days prior to standard of care conditioning chemotherapy and continuing until discharge from the hospital. Stool will be collected at different time points throughout the study. Patients may also undergo blood sample collection throughout the study.
  Interventions: Other: Survey Administration; Dietary Supplement: Dietary Supplement; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Fiber and Dietary Assessments

INTERVENTIONS:
Dietary Supplement: Kate Farms 1.0 — Given enteral nutrition via nasoenteric feeding
  Other Names: Polymeric Enteral Nutrition Formula
  Arms: Arm I (enteral nutrition) [Discontinued in January 2024]
Dietary Supplement: Standard of Care Nutritional Support — Given standard of care, which may be parenteral nutrition
  Other Names: hyperalimentation; parenteral nutrition; Total Parenteral Nutrition; TPN
  Arms: Arm II (standard of care) [Discontinued in January 2024]
Other: Survey Administration — Ancillary studies
Dietary Supplement: Dietary Supplement — Receive fiber supplementation orally or enterally
  Other Names: nutritional supplement; supplemental nutrition; Supplements
  Arms: Supportive care (Fiber) [Current study activity]
Procedure: Biospecimen Collection — Undergo collection of blood and stool samples
  Arms: Supportive care (Fiber) [Current study activity]
Other: Electronic Health Record Review — Ancillary studies
  Arms: Supportive care (Fiber) [Current study activity]
Other: Fiber and Dietary Assessments — Ancillary studies
  Arms: Supportive care (Fiber) [Current study activity]

SUMMARY:
This clinical trial examines sustained oral fiber supplementation for patients undergoing donor stem cell transplantation for hematological malignancies. Patients undergoing donor stem cell transplantation often develop oral and gastrointestinal damage from chemotherapy, radiotherapy, or graft-versus-host disease. Oral fiber nutrition support may improve overall nutrition, support a normal gut microbiome (bacteria that live in the gut) and/or improve gut function in patients undergoing stem cell transplants.

DETAILED DESCRIPTION:
OUTLINE:

Current study design: Patients receive fiber supplementation orally (PO) or enterally starting 14 to 5 days prior to standard of care conditioning chemotherapy and continuing until discharge. Patients who are not able to receive sufficient nutrition by mouth may receive parenteral nutrition or enteral nutrition by feeding tube from the hospital. Patients may undergo blood sample collection throughout the study.

Previous study design: Before this study was amended in January 2024, patients were randomized to 1 of 2 arms.

Previous Arm I: Patients received enteral nutrition via nasoenteric feeding tube starting on day 1 until hospital discharge.

Previous Arm II: Patients received standard of care nutritional support.

After completion of study treatment, patients are followed up at days 42, 60 and 90 days post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to initiation of any study procedures
* Planned allogeneic stem cell transplantation
* At least 18 years of age

Exclusion Criteria:

* Major psychiatric diagnosis that impairs cognitive functioning or is not controlled at the time of the approach, as judged by the patient's medical team
* Pregnant or breastfeeding. Pregnancy test is obtained as part of pre-transplant evaluation in women of child-bearing potential at arrival to transplant and again within 7 days of conditioning and will be confirmed as negative by review of the chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Study participation rates | Assessed at consenting
  The proportion of eligible patients who consent to enroll in the study will be computed based on the number approached and estimated with 95% confidence intervals.

SECONDARY OUTCOMES:
Number of days receiving at least 10 grams of fiber | Up to 90 days following transplant
Number of days receiving at least 25 grams of fiber | Up to 90 days following transplant
Tolerance of initiating and maintaining oral fiber intake | Up to 90 days following transplant
  Tolerance of initiating and maintaining oral fiber intake (or via enteral nutrition) will be calculated as delivery of the intended amount on each day that nutritional supplementation was indicated.
Level of comfort/distress attributed to initiating and maintaining oral fiber intake | Up to 90 days following transplant
  The post-discharge questions measuring level of comfort or distress experienced with each nutritional treatment will be tabulated.
Incidence of adverse events | Up to 90 days following transplant
  Will assess safety including diarrhea, abdominal pain, bloating.

CONTACTS AND LOCATIONS:
Overall Officials: David Fredricks, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No